CLINICAL TRIAL: NCT04120792
Title: The Aerobic and Cognitive Training System to Improve Cognition
Brief Title: The Aerobic and Cognitive Training System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UA15-011
Record Dates: First submitted 2019-10-04; First posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-05

CONDITIONS: Healthy Aging
MeSH Terms: interventions — Cognitive Training; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (4):
- Simultaneous exercise and cognitive training (Experimental): Participants in this arm will engage in a 12-week intervention that combines physical exercise and cognitive tablet-based training. This intervention involves use of an exercise bicycle while engaging in cognitive tasks on a tablet computer three times per week.
  Interventions: Behavioral: Simultaneous exercise and cognitive training
- Exercise training (Active Comparator): Participants in this arm will engage in a 12-week exercise intervention that involves use of an exercise bicycle three times per week.
  Interventions: Behavioral: Exercise training
- Cognitive training (Active Comparator): Participants in this arm will engage in a 12-week intervention that involves cognitive tablet-based training three times per week.
  Interventions: Behavioral: Cognitive Training
- Neutral Video (Active Comparator): Participants in this arm will engage in a 12-week intervention that involves watching neutral videos on a tablet computer three times per week.
  Interventions: Behavioral: Neutral video

INTERVENTIONS:
Behavioral: Simultaneous exercise and cognitive training — Participants in this arm will engage in a 12-week intervention that combines physical exercise and cognitive tablet-based training. This intervention involves use of an exercise bicycle while engaging in cognitive tasks on a tablet computer three times per week.
  Arms: Simultaneous exercise and cognitive training
Behavioral: Exercise training — Participants in this arm will engage in a 12-week exercise intervention that involves use of an exercise bicycle three times per week.
  Arms: Exercise training
Behavioral: Cognitive Training — Participants in this arm will engage in a 12-week intervention that involves cognitive tablet-based training three times per week.
  Arms: Cognitive training
Behavioral: Neutral video — Participants in this arm will engage in a 12-week intervention that involves watching neutral videos on a tablet computer three times per week.
  Arms: Neutral Video

SUMMARY:
This study will determine the effects of simultaneous exercise and cognitive training on cognitive function in healthy older adults. Specifically, this study will compare the use of a tablet-based cognitive training system while exercising with exercise alone, cognitive training alone, and a neutral control condition on cognition.

ELIGIBILITY:
Inclusion Criteria:

Generally healthy, age 60-74, and a written statement from their primary care physician indicating that they are able to participate in the 12-week exercise program.

Exclusion Criteria:

Subjects will be excluded from participating in the study if they express significant concerns about their memory or declines in other cognitive abilities, if they are not English speaking, or if they have histories of significant major neurological, psychiatric, or medical disorder or injury that would affect cognitive function.

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cognitive function during dual-task test at 12 weeks | Baseline and 12-weeks
  Performance on serial subtraction during dual-task walking.

SECONDARY OUTCOMES:
Change from baseline in stride length during dual-task test | Baseline, 6 weeks, 12 weeks
  The difference between stride length in single and dual-task walking will be assessed at baseline, 6 weeks, and 12 weeks
Change from baseline in stride duration during dual-task test | Baseline, 6 weeks, 12 weeks
  The difference between stride duration in single and dual-task walking will be assessed at baseline, 6 weeks, and 12 weeks
Change from baseline in stride velocity during dual-task test | Baseline, 6 weeks, 12 weeks
  The difference between stride velocity in single and dual-task walking will be assessed at baseline, 6 weeks, and 12 weeks
Change from baseline in stride length variability during dual-task test | Baseline, 6 weeks, 12 weeks
  The difference between stride length variability (measured by coefficient of variation) in single and dual-task walking will be assessed at baseline, 6 weeks, and 12 weeks
Change from baseline in stride duration variability during dual-task test | Baseline, 6 weeks, 12 weeks
  The difference between stride duration variability (measured by coefficient of variation) in single and dual-task walking will be assessed at baseline, 6 weeks, and 12 weeks
Change from baseline in stride velocity variability during dual-task test | Baseline, 6 weeks, 12 weeks
  The difference between stride velocity variability (measured by coefficient of variation) in single and dual-task walking will be assessed at baseline, 6 weeks, and 12 weeks
Change from baseline in cognitive function during dual-task test at 6 weeks | Baseline and 6-weeks
  Performance on serial subtraction during dual-task walking.

OTHER OUTCOMES:
Change from baseline in Wechsler Adult Intelligence Scale-IV Digit Span total score | Baseline, 6 weeks, 12 weeks
  A measure of working memory
Change from baseline in Wechsler Adult Intelligence Scale-IV Coding total score | Baseline, 6 weeks, 12 weeks
  A measure of information processing
Change from baseline in Wechsler Adult Intelligence Scale-IV Letter-Number Sequencing total score | Baseline, 6 weeks, 12 weeks
  A measure of working memory
Change from baseline in Wechsler Memory Scale-IV Paired-Associates I total score | Baseline, 6 weeks, 12 weeks
  A measure of verbal learning
Change from baseline in Auditory Verbal Learning Test total learning score | Baseline, 6 weeks, 12 weeks
  A test of verbal list learning
Change from baseline in Trail Making Test, part A total time | Baseline, 6 weeks, 12 weeks
  Tests of visuomotor tracking and complex attention
Change from baseline in Trail Making Test, part B total time | Baseline, 6 weeks, 12 weeks
  Tests of visuomotor tracking and complex attention
Change from baseline in Stroop Color and Word Test Color/Word Interference total score | Baseline, 6 weeks, 12 weeks
  A test to assess inhibition when reading color words
Change from baseline in Deary-Liewald Reaction Time Task Simple median response time | Baseline, 6 weeks, 12 weeks
  Tests to measure speed of information processing
Change from baseline in Deary-Liewald Reaction Time Task Choice median correct response time | Baseline, 6 weeks, 12 weeks
  Tests to measure speed of information processing

CONTACTS AND LOCATIONS:
Overall Officials: Gene Alexander, Principal Investigator — University of Arizona; David Raichlen, Principal Investigator — University of Arizona

REFERENCES:
- [Derived] Raichlen DA, Bharadwaj PK, Nguyen LA, Franchetti MK, Zigman EK, Solorio AR, Alexander GE. Effects of simultaneous cognitive and aerobic exercise training on dual-task walking performance in healthy older adults: results from a pilot randomized controlled trial. BMC Geriatr. 2020 Mar 2;20(1):83. doi: 10.1186/s12877-020-1484-5. PMID 32122325